CLINICAL TRIAL: NCT01037270
Title: Evaluation of the Accuracy and Precision of the INRatio® Prothrombin Time (PT) Monitoring System With New INRatio Test Strip Designed for Low Sample Volume and Heparin Insensitivity
Acronym: ECLIPSE-01
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Sponsor
Other Study IDs: BSTE-0124
Record Dates: First submitted 2009-12-17; First posted 2009-12-22 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Pulmonary Embolism; Atrial Fibrillation; Deep Vein Thrombosis
Keywords: Patients with conditions (PE, Afib, DVT) requiring ongoing INR measurements.
MeSH Terms: conditions — Pulmonary Embolism; Atrial Fibrillation; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma specimens for reference testing.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center study designed to evaluate the accuracy and precision of the INRatio® Prothrombin Time (PT) Monitoring System, utilizing the INRatio test strip newly designed for low sample volume and heparin insensitivity, when used by trained medical professionals for the quantitative determination of PT and International Normalized Ratio (INR) in fingerstick and venous whole blood from subjects on oral anticoagulation therapy (OAT). These results will be compared to those PT/INR results obtained on plasma from the same subjects as analyzed at a central laboratory with the Sysmex CA-560 System.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older);
* Willing and able to provide written informed consent and comply with study procedures;
* Subjects on oral anticoagulation therapy. This inclusion criterion is waived for the 20 normal healthy volunteers who must NOT be on warfarin or any other anticoagulant drug.

Exclusion Criteria:

* Hematocrit less than 25 or greater than 55%;
* Lupus or antiphospholipid syndrome (APS)
* Vulnerable populations deemed inappropriate for study by the site's principal investigator.
* Already participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 210 subjects on OAT and 20 normal healthy subjects not on anticoagulation therapy will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Analytical accuracy and precision of the INRatio Prothrombin Time (PT) Monitoring System. | 3-6 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Loma Linda VA Hospital, Loma Linda, California
  - UC Davis Healthcare System, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - Fox Valley Cardiology, Aurora, Illinois